CLINICAL TRIAL: NCT00541554
Title: Reversal of Antipsychotic-Induced Hyperprolactinemia, Weight Gain, Hyperglycemia and Dyslipidemia by Aripiprazole Add-on Therapy in the Treatment of Schizophrenia and Bipolar Disorder: An Open-Label Trial
Brief Title: Reversal of Antipsychotic-Induced Hyperprolactinemia, Weight Gain, Hyperglycemia and Dyslipidemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genovate Biotechnology Co., Ltd., (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-06-P05
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Hyperprolactinemia; Weight Gain; Dyslipidemia
MeSH Terms: conditions — Hyperprolactinemia; Weight Gain; Dyslipidemias | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Abilify (aripiprazole)

SUMMARY:
This is a prospective, open-label study to evaluate the efficacy and safety in reducing antipsychotic-induced hyperprolactinemia, weight gain, and dyslipidemia by aripiprazole. Approximate 60 patients will be recruited to achieve at least 40 evaluable patients.

DETAILED DESCRIPTION:
A.Screening / Baseline visit (V1; Day 0) After signing the informed consent form, patients' DSM-IV multiaxial examination, physical examination, vital sign, pregnancy test, BMI will be conducted. The demographics, medical history, and concomitant medication will be recorded. After evaluating all variables obtained, the eligible patients will be enrolled into study.Patients who fulfill the inclusion / exclusion criteria will be performed the laboratory tests, PANSS, EPS (AIMS & BARS), menstrual function, sexual function (Arizona sexual experience scale) and prolaction. Afterwards, the treatment period will be started to add-on with first medication (7.5 or 15 mg daily by patient, which was prescribed by investigator) to current antipsychotics at this visit. Besides, drug accounting and adverse events will also be recorded at this visit. Patients are maintained on current doses of antipsychotics, and all other medicines.

B.Treatment phase (V2~V3; 2~4 Week finished; 14±3~28±3 Day finished) The vital sign, physical examination, BMI, laboratory tests (at V3), PANSS, EPS (AIMS & BARS), menstrual function, sexual function (Arizona sexual experience scale), and prolactin will be carried out. Concomitant medication, adverse events, and drug accounting will also be recorded at this visit. Study drug could be titrated with a flexible dose from 7.5 to 30 mg QD. All dose adjustments should be made with the approval of the investigator.

C.Completion visit (V4; 8 Week Finished; 56±7 Day finished, or Early termination) The vital sign, physical examination, pregnancy test, BMI, laboratory tests, PANSS, EPS (AIMS & BARS), menstrual function, sexual function (Arizona sexual experience scale), prolactin will be carried out. Concomitant medication, adverse events, and drug accounting will also be recorded at this visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in age between 12 and 65 years old.
2. Clinical diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder with DSM-IV criteria.
3. Keep stable dosage of the same antipsychotic other than aripiprazole during last one month.
4. Who are currently taking antipsychotic drugs and for whom an alteration in medication is clinically reasonable. This includes patients who are stable or who have symptoms that are not optimally controlled or patients experiencing tolerability problems.
5. Having antipsychotic-induced symptomatic hyperprolactinemia, weight gain, increased plasma glucose or dyslipidemia judged by the investigator.
6. Informed Consent was obtained from the subject and legal guardian (if necessary).

Exclusion Criteria:

1. Pregnant or breast feeding women or planning a pregnancy.
2. Patient has a history of hypersensitivity or allergy to investigated drug.
3. Acute psychosis, acute suicidal ideation, or any acute psychiatric condition that might require emergent intervention.
4. Any clinical condition or significant concurrent disease judged by the investigator to complicate the evaluation of the study treatment.
5. Having participated other investigational drug study and taken the investigation drug within one month prior to study entry.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-10; Study Completion 2009-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Chih-Ken, PhD, Principal Investigator — Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Derived] Chen CK, Huang YS, Ree SC, Hsiao CC. Differential add-on effects of aripiprazole in resolving hyperprolactinemia induced by risperidone in comparison to benzamide antipsychotics. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Dec 1;34(8):1495-9. doi: 10.1016/j.pnpbp.2010.08.012. Epub 2010 Aug 20. PMID 20732372